CLINICAL TRIAL: NCT07396883
Title: Developmental and Epileptic Encephalopathies Diagnosed Via Long-read Genome Sequencing - EEPILOG
Brief Title: Developmental and Epileptic Encephalopathies Diagnosed Via Long-read Genome Sequencing
Acronym: EEPILOG
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: IGBMC (Unknown); Laboratoire de diagnostic génétique - NHC (Unknown); Groupe Méthode en Recherche Clinique (GMRC) (Unknown); Bio-informatique médicale appliquée au diagnostic (UF7363) - NHC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 9964
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Developmental and Epileptic Encephalopathy; Epilepsy in Children
Keywords: Developmental and Epileptic Encephalopathy (DEE); Drug-Resistant Epilepsy; Long-read Whole Genome Sequencing (lrWGS); Long-read Sequencing; Negative Short-read Sequencing; Genetic Diagnosis; Pediatric Neurology; High-Throughput Nucleotide Sequencing; Early-Onset Epilepsy; Genetic Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DEE Long-read: his cohort is composed of pediatric patients (under 18 years old) with Developmental and Epileptic Encephalopathy (DEE) as defined by the 2022 ILAE criteria.
  The group is specifically characterized by a prior negative molecular diagnosis despite analysis via short-read Whole Genome Sequencing (srWGS) through the French Genomic Medicine Plan 2025 (AURAGEN platform).
  Selection follows a clinical prioritization strategy: while the study includes all eligible DEE patients without a genetic answer, priority is given to those with early-onset forms, familial cases, or current therapeutic impasse (patients for whom standard treatments have failed). The study excludes cases where a clear non-genetic cause is identified, such as perinatal brain injury, focusing the cohort on high-probability "hidden" genetic etiologies.
  Interventions: Diagnostic Test: Long-read Whole Genome Sequencing (lrWGS)

INTERVENTIONS:
Diagnostic Test: Long-read Whole Genome Sequencing (lrWGS) — Long-read Whole Genome Sequencing (lrWGS) using high-molecular-weight DNA previously extracted and banked during the patient's initial clinical workup.

SUMMARY:
This study focuses on children with Developmental and Epileptic Encephalopathy (DEE), a severe form of epilepsy that often has a genetic origin. Currently, standard diagnostic tools-known as short-read genome sequencing-fail to provide a diagnosis for over 50% of affected patients because they cannot detect certain complex DNA abnormalities.

The purpose of this study is to evaluate the effectiveness of a newer, more advanced technology called Long-read Genome Sequencing (lrWGS). Unlike traditional methods, this technology analyzes very long fragments of DNA, allowing researchers to identify genetic errors that were previously "invisible."

The study aims to answer whether Long-read Sequencing can successfully identify the genetic cause of epilepsy in patients who have already received a negative result from standard testing. By finding these missing answers, the research seeks to enable personalized medical treatments, improve genetic counseling for families, and advance our understanding of how these complex neurological conditions develop.

DETAILED DESCRIPTION:
This study evaluates the clinical utility of Long-read Whole Genome Sequencing (lrWGS) as a secondary diagnostic tool for Developmental and Epileptic Encephalopathies (DEEs). While current standard-of-care "short-read" sequencing (srWGS) is effective at identifying small genetic mutations, it often fails to detect complex structural changes, leaving over 50% of patients without a diagnosis.

Technically, lrWGS overcomes these limitations by analyzing DNA fragments that are thousands of bases long. This allows researchers to map "dark regions" of the genome and identify Structural Variants (SVs), such as large insertions, deletions, or repeat expansions, which are often the hidden causes of severe epilepsy.

By identifying these elusive genetic drivers, the study aims to move beyond a simple diagnosis toward precision medicine. A clear molecular result can directly influence clinical decisions, such as selecting targeted medications, avoiding contraindicated drugs, or determining eligibility for emerging gene therapies. Additionally, the project assesses the feasibility of integrating this technology into routine clinical practice by evaluating bioinformatic complexity and diagnostic turnaround times.

ELIGIBILITY:
Inclusion Criteria:

Pediatric Participants:

* Age < 18 years.
* Diagnosis of Developmental and Epileptic Encephalopathy (DEE) according to 2022 ILAE criteria (severe epilepsy, encephalopathic EEG, multiple drug-resistant seizures, and neurodevelopmental disorder).
* Brain MRI without markers of perinatal anoxia.
* Negative molecular diagnosis after short-read Whole Genome Sequencing (srWGS) via the French Genomic Medicine Plan 2025 (AURAGEN).
* Available banked DNA at a participating center.

Parents/Legal Guardians:

* Age ≥ 18 years.
* Able to understand study objectives and risks.
* Signed and dated informed consent.
* Affiliated with or beneficiary of a social security scheme.

Exclusion Criteria:

Pediatric Participants:

* Brain MRI findings in favor of perinatal cerebral anoxia.
* Intercurrent diseases preventing the completion of protocol examinations.
* Subject currently in an exclusion period from another study.

Parents/Legal Guardians:

* Inability to receive or understand informed information (e.g., life-threatening emergency).
* Subject under judicial protection, tutelage, or curatorship.
* Language barriers where an official interpreter is unavailable.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is drawn from specialized pediatric neurology and genetics departments within the French university hospital network (CHU).
  Participants are specifically sourced from the existing patient base of the AURAGEN platform, one of the two national sequencing hubs established under the French Genomic Medicine Plan 2025 (PFMG 2025). These individuals represent a highly selected sub-population of children across France who have already undergone extensive clinical phenotyping and "first-line" genomic screening but remain without a molecular diagnosis.
  The recruitment occurs primarily at the Strasbourg University Hospital (Hôpitaux Universitaires de Strasbourg) and collaborating clinical sites. These centers serve as regional and national referral points for rare and refractory childhood epilepsies, ensuring that the study population includes the most complex and diagnostically challenging cases of Developmental and Epileptic Encephalopathy (DEE) in the country.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of pathogenic and likely pathogenic genetic variants identified by long-read whole genome sequencing (lrWGS) | At the results delivery visit (Visit 1), up to 15 months after enrollment.
  Evaluate the efficacy of long-read whole genome sequencing (lrWGS) in identifying genetic causes in patients with developmental and epileptic encephalopathy who did not obtain a molecular diagnosis despite previous short-read whole genome sequencing (srWGS) analysis within the framework of the French Genomic Medicine Plan 2025 (PFMG 2025).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Jean Minjoz, Besançon
  - American Memorial Hospital, Reims
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Nancy - hôpital d'enfant, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No